CLINICAL TRIAL: NCT05821855
Title: A Postmarketing Study Evaluating the Effectiveness and Safety of the XEN45 Glaucoma Treatment System in Subjects With Open-Angle Glaucoma in China
Brief Title: A Study to Evaluate Adverse Events and Change in Disease Activity With the XEN45 Glaucoma Treatment System Implantation In Adult Participants With Open-Angle Glaucoma in China
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1924-802-007
Record Dates: First submitted 2023-03-23; First posted 2023-04-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Open-angle Glaucoma; OAG
Keywords: Open-angle glaucoma; OAG; XEN45; Intraocular pressure; IOP
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- XEN45 (Experimental): Participants will be implanted with the XEN45 glaucoma treatment system in the study eye on Day 1 and followed for 60 months.
  Interventions: Device: XEN45 Glaucoma Treatment System
- Trabeculectomy (Active Comparator): Participants will undergo trabeculectomy in the study eye on Day 1 and followed for 60 months.
  Interventions: Procedure: Trabeculectomy

INTERVENTIONS:
Device: XEN45 Glaucoma Treatment System — Ab interno implantation
  Arms: XEN45
Procedure: Trabeculectomy — Surgical Intervention
  Arms: Trabeculectomy

SUMMARY:
Glaucoma is the second most common cause of blindness in the world, second only to cataracts. The purpose of this study is to assess adverse events (AEs) and changes in disease activity in participants with open-angle glaucoma (OAG) receiving the XEN45 Glaucoma Treatment System (XEN45).

XEN45 is an approved device for the treatment of OAG in participants in China who have not achieved satisfactory effectiveness with or are not suitable for intraocular pressure (IOP)-lowering medication, laser surgery, or are not tolerant of traditional filtration surgery. Adult participants with a diagnosis of OAG will be randomized to receive either XEN 45 or trabeculectomy. Around 130 participants will be enrolled in the study at approximately 15 sites in China.

Participants will receive XEN45 implanted using the ab interno approach or trabeculectomy on Day 1 and will be followed for 60 months

An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Area of healthy, free, and mobile conjunctiva in the target area in the study eye, i.e., superior bulbar conjunctiva.
* Visible trabecular meshwork with Shaffer angle grade => 3 in the study eye at the Screening Visit.
* IOP => 20 mm Hg and <= 44 mm Hg for the study eye, measured by Goldmann applanation tonometer, at the Screening Visit and Baseline Visit.

Exclusion Criteria:

* Active neovascular, uveitic, or angle-recession glaucoma or any glaucoma-associated vascular disorders within 6 months of the Screening Visit in the study eye.
* Prior XEN45, transscleral cycloablative procedures (such as cyclophotocoagulation, micropulse cyclophotocoagulation, cryotherapy, ultrasonic circular cyclocoagulation [UC3], etc.) or prior major conjunctival surgery (i.e., scleral buckle) in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Intraocular Pressure (IOP) | Baseline to Month 12
  IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Number of Participants with Adverse Events (AEs) | Baseline to Month 60
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants with Treatment Response of Achieving => 20% IOP Reduction | Baseline to Month 12
  Treatment response is defined as IOP reduction on the same or fewer number of topical IOP-lowering medications without secondary surgical intervention (SSI) for uncontrolled IOP.
Change from Baseline in IOP by Visit | Baseline to Month 12
  IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Change from Baseline in Number of Topical IOP-Lowering Medications | Baseline to Month 12
  A numerical count by class of drug of topical IOP lowering medications being taken.
Percentage of Participants Achieving IOP <= 18 mm Hg and => 20% mean IOP reduction from Baseline Without Topical IOP-lowering Medications | Baseline to Month 12
  The complete treatment response is defined as the percentage of participants achieving IOP <=18 mm Hg and 20% or more reduction of IOP without topical IOP medications from baseline.
Percentage of Participants Achieving IOP <= 18 mm Hg and => 20% mean IOP Reduction from Baseline With Any Topical IOP-Lowering Medications | Baseline to Month 12
  The qualified treatment response is defined as the percentage of participants achieving IOP <= 18 mm Hg and 20% mean IOP reduction from baseline with any topical IOP-lowering medications.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (13):
- China (13):
  - Peking University people s hospital /ID# 265493, Beijing, Beijing Municipality
  - Peking University Third Hospital /ID# 243994, Beijing, Beijing Municipality
  - Beijing Tongren Hospital Affiliated To Capital Medical University /ID# 244055, Beijing, Beijing Municipality
  - The First Affiliated Hospital Of Fujian Medical University /ID# 244004, Fuzhou, Fujian
  - Xiamen Eye Center of Xiamen University /ID# 244000, Xiamen, Fujian
  - The Second Affiliated Hospital of Guangzhou Medical University /ID# 275493, Guangzhou, Guangdong
  - Shenzhen Eye Hospital /ID# 244001, Shenzhen, Guangdong
  - Tongji Hospital Tongji Medical College of HUST /ID# 243998, Wuhan, Hubei
  - Qingdao Eye Hospital Of Shandong First Medical University /ID# 243992, Qingdao, Shandong
  - West China Hospital, Sichuan University /ID# 243999, Chengdu, Sichuan
  - Tianjin Eye Hospital /ID# 243997, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine /ID# 243996, Hangzhou, Zhejiang
  - Zhongshan Ophthalmic Center,SunYat-Sen University /ID# 243843, Guangzhou

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — http://www.abbvieclinicaltrials.com/study/?id=1924-802-007